CLINICAL TRIAL: NCT01838889
Title: Exploratory RCT of a Group Psychological Intervention for Postnatal Depression in British Mother's of South Asian Origin
Brief Title: Exploratory Trial of a Group Psychological Intervention for Postnatal Depression in British Mother's of South Asian Origin
Acronym: ROSHNI-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancashire Care NHS Foundation Trust (Network)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 47847; PB-PG-1208-18087 (Other Grant/Funding Number: NIHR Research for Patient Benefit)
Record Dates: First submitted 2013-04-14; First posted 2013-04-24 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Depression, Postpartum; Postnatal Depression in British South Asian Women
Keywords: Culturally adapted; Group psychological intervention; British South Asian women; CBT
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Culturally adapted psychological intervention (PHP) (Experimental): Depressed Mothers randomized to experimental arm will undergo a 12 week group psychological intervention on the 'positive health programme'.
  Interventions: Behavioral: Culturally adapted psychological intervention (Positive Health Programme)
- Treatment as usual (TAU) (No Intervention): Depressed mothers randomized to TAU arm will receive treatment as usual.

INTERVENTIONS:
Behavioral: Culturally adapted psychological intervention (Positive Health Programme) — This study will evaluate the efficacy of a group psychological intervention (PHP) based on the principles of Cognitive Behaviour Therapy in treating depression in postpartum women.
  Other Names: PHP
  Arms: Culturally adapted psychological intervention (PHP)

SUMMARY:
This study is an exploratory randomized controlled trial (RCT) of a group psychological intervention for postnatal depression in British mother's of south Asian origin. The aim is to evaluate the efficacy of a group psychological intervention (PHP) based on the principles of Cognitive Behaviour Therapy in treating depression in postpartum women. The hypothesis is that depressed British women of South Asian origin receiving the group intervention will show significant improvements in terms of severity of depression as compared to the treatment as usual (TAU) control group.

ELIGIBILITY:
Inclusion Criteria:

* self-ascribed British women of South Asian origin as defined by UK Office of -National Statistics,
* over the age of 16 years
* living with their babies,
* who meet the criteria for ICD-10 depression

Exclusion Criteria:

* women with diagnosed physical or learning disability,
* post-partum or other psychosis,
* severely depressed
* actively suicidal.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Edinburgh Post Natal Depression Scale (EPDS; Cox et al 1987) | Assessments will be carried out at baseline, 3 months (end of intervention) and 6 months (The primary end point is 3 months).

SECONDARY OUTCOMES:
EuroQoL-5 Dimensions (EQ-5D) | Assessments will be carried out at baseline, 3 months (end of intervention) and 6 months (The primary end point is 3 months)
The Parenting Stress Index (PSI) | Assessments will be carried out at baseline, 3 months (end of intervention) and 6 months (The primary end point is 3 months)
Multidimensional Scale of Perceived Social Support (MSPSS) | Assessments will be carried out at baseline, 3 months (end of intervention) and 6 months (The primary end point is 3 months)
Dyadic Adjustment Scale (DAS) | Assessments will be carried out at baseline, 3 months (end of intervention) and 6 months (The primary end point is 3 months)
Home Inventory (HI) | Assessments will be carried out at baseline, 3 months (end of intervention) and 6 months (The primary end point is 3 months)
Hamilton Rating Scale for Depression (HRSD) | Assessments will be carried out at baseline, 3 months (end of intervention) and 6 months (The primary end point is 3 months)
Client Service Receipt Inventory (CSRI) | Assessments will be carried out at baseline, 3 months (end of intervention) and 6 months (The primary end point is 3 months)

OTHER OUTCOMES:
Revised Clinical Interview Schedule (CIS-R) | Assessment done at baseline
  Tool used to confirm the diagnosis of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care; Mother and Baby Clinics, Borough of Blackburn With Darwen; Burnley; Preston; Manchester, Lancashire, Greater Manchester, United Kingdom

REFERENCES:
- [Derived] Husain N, Lunat F, Lovell K, Sharma D, Zaidi N, Bokhari A, Syed A, Tomenson B, Islam A, Chaudhry N, Waheed W. Exploratory RCT of a group psychological intervention for postnatal depression in British mothers of South Asian origin - ROSHNI-D. Acta Psychol (Amst). 2023 Aug;238:103974. doi: 10.1016/j.actpsy.2023.103974. Epub 2023 Jul 4. PMID 37413896
- [Derived] Masood Y, Lovell K, Lunat F, Atif N, Waheed W, Rahman A, Mossabir R, Chaudhry N, Husain N. Group psychological intervention for postnatal depression: a nested qualitative study with British South Asian women. BMC Womens Health. 2015 Nov 25;15:109. doi: 10.1186/s12905-015-0263-5. PMID 26603604